CLINICAL TRIAL: NCT02259725
Title: Phase II Study of Single Agent Regorafenib in Patients With Advanced/Metastatic Neuroendocrine Tumors
Brief Title: Regorafenib in Treating Patients With Advanced or Metastatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0S-14-3; NCI-2014-01996 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-14-00583; 0S-14-3 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Gastrinoma; Glucagonoma; Insulinoma; Metastatic Gastrointestinal Carcinoid Tumor; Pancreatic Polypeptide Tumor; Pulmonary Carcinoid Tumor; Recurrent Gastrointestinal Carcinoid Tumor; Recurrent Islet Cell Carcinoma; Somatostatinoma
MeSH Terms: conditions — Gastrinoma; Glucagonoma; Insulinoma; Carcinoma, Islet Cell; Somatostatinoma | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (regorafenib) (Experimental): Patients receive regorafenib PO QD on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: regorafenib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: regorafenib — Given PO
  Other Names: BAY 73-4506; multikinase inhibitor BAY 73-4506; Stivarga
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies regorafenib in treating patients with neuroendocrine tumors that have spread from the primary site (place where it started) to other places in the body. Regorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess progression-free survival (PFS) in advanced/metastatic in patients with carcinoid or pancreatic islet cell tumors.

SECONDARY OBJECTIVES:

I. To assess overall survival and response rate in advanced/metastatic poor prognosis in patients with carcinoid or pancreatic islet cell tumors.

II. To assess the toxicity of patients treated with regorafenib. III. To explore markers of angiogenesis as they relate to outcome in carcinoid and pancreatic islet cell tumors.

OUTLINE:

Patients receive regorafenib orally (PO) once daily (QD) on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Advanced metastatic, progressing carcinoid or pancreatic islet cell cancers
* No prior targeted treatment (tx) or anti-angiogenic therapy; patients may have received one line of prior therapy with octreotide, locoregional therapy; continuation of concurrent octreotide is allowed; patients will be maintained on octreotide (sandostatin) for the duration of their treatment
* Life expectancy of at least 12 weeks (3 months)
* Subjects must be able to understand and be willing to sign the written informed consent form (ICF); a signed ICF must be appropriately obtained prior to the conduct of any trial-specific procedure
* All acute toxic effects of any prior treatment have resolved to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version (v)4.0 grade 1 or less at the time of signing the informed consent form (ICF); exceptions to this include alopecia
* Total bilirubin =< 1.5 x the upper limits of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer)
* Alkaline phosphastase limit =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer)
* Lipase =< 1.5 x the ULN
* Amylase =< 1.5 x the ULN
* Serum creatinine =< 1.5 x the ULN
* International normalized ratio (INR)/ partial thromboplastin time (PTT) < 1.5 x ULN; (subjects who are treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists; close monitoring [day 5 of cycle 1 and day 1 of each cycle] is mandatory) will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care)
* Platelet count >= 100,000 /mm^3
* Hemoglobin (Hb) >= 9 g/dL
* Absolute neutrophil count (ANC) >= 1,500/mm^3; blood transfusion to meet the inclusion criteria will not be allowed
* Glomerular filtration rate (GFR) >= 30 ml/min/1.73 m^2 according to the Modified Diet in Renal Disease (MDRD) abbreviated formula
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug; post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test; the definition of adequate contraception will be based on the judgement of the investigator
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 3 months after the last dose of study drug; the definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate
* Subject must be able to swallow and retain oral medication
* Southwest Oncology Group (SWOG) performance status 0-1
* Patients must have measurable disease

Exclusion Criteria:

* Previous assignment to treatment during this study; subjects permanently withdrawn from study participation will not be allowed to re-enter study
* Uncontrolled hypertension (systolic pressure > 140 mm Hg or diastolic pressure > 90 mm Hg [NCI-CTCAE v4.0] on repeated measurement) despite optimal medical management
* Active or clinically significant cardiac disease including:

  * Congestive heart failure - New York Heart Association (NYHA) > class II
  * Active coronary artery disease
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin
  * Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization
* Evidence or history of bleeding diathesis or coagulopathy
* Any hemorrhage or bleeding event >= NCI-CTCAE grade 3 within 4 weeks prior to start of study medication
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of start of study treatment
* Subjects with any previously untreated or concurrent cancer that is distinct in primary site or histology from carcinoid or pancreatic islet cancer except cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor; subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before randomization are allowed; all cancer treatments must be completed at least 3 years prior to study entry (i.e., signature date of the informed consent form)
* Patients with pheochromocytoma
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy
* Ongoing infection > grade 2 NCI-CTCAE v4.0
* Presence of a non-healing wound, non-healing ulcer, or bone fracture
* Renal failure requiring hemo-or peritoneal dialysis
* Dehydration grade >= 1 NCI-CTCAE v4.0
* Patients with seizure disorder requiring medication
* Persistent proteinuria >= grade 3 NCI-CTCAE v4.0 (> 3.5 g/24 hrs, measured by urine protein:creatinine ratio on a random urine sample)
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
* Pleural effusion or ascites that causes respiratory compromise (>= NCI-CTCAE version 4.0 grade 2 dyspnea)
* History of organ allograft (including corneal transplant)
* Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial
* Any malabsorption condition
* Women who are pregnant or breast-feeding
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to regorafenib or other agents used in study
* Uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Excluded therapies and medications, previous and concomitant

  * Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) other than study treatment (regorafenib)
  * Prior use of regorafenib
  * Concurrent use of chemotherapy, radiotherapy or another investigational drug or device therapy (i.e., outside of study treatment) during, or within 4 weeks of trial entry (signing of the ICF)
  * Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication
  * Use of any herbal remedy (e.g. St. John's wort [Hypericum perforatum])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, MD, Principal Investigator — University of Southern California
Locations (5):
- United States (5):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - USC Norris Oncology Hematology-Newport Beach, Newport Beach, California
  - Seattle Cancer Care Alliance, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began recruiting in August 2016 and ended in January 2019. All subjects were seen and treated either at USC Norris Comprehensive Cancer Center or at LAC+USC Medical Center.
Pre-assignment Details: There were no pre-assignment criteria. All subjects were given the same treatment.
Period: Overall Study
Arm/Group | Treatment (Regorafenib)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Regorafenib)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: PFS
Description: Two parallel Simon's 2-stage phase II trials will be conducted to evaluate the efficacy of regorafenib in patients with advanced carcinoid (cohort A) or pancreatic islet cell tumors (cohort B). Will be summarized as a proportion of patients who are alive and progression-free among all patients in the primary data analysis set. The 95% confidence intervals (CIs) will be calculated using the Wilson method. Will be analyzed using Kaplan-Meier (KM) curves. The median PFS and 95% CIs will be calculated. The probability of 6-month PFS will be estimated from the KM curve too.
Time Frame: Time from start of treatment to time of progression or death on study whichever comes first, assessed at 6 months
Population: No analysis done. Only 3 subjects were enrolled out of accrual goal of 24 subjects.
Arm/Group | Treatment (Regorafenib)
Number analyzed (Participants) | 0

2. Secondary Outcome: Tumor Response Rate, Evaluated Using the New International Criteria Proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee
Description: Will be calculated as a proportion of patients who have either a complete or partial response among all patients in the primary data analysis set. The 95% CIs will be given.
Time Frame: Up to 4 years
Population: No analysis was done. Only 3 subjects were enrolled out of accrual goal of 24 subjects.
Arm/Group | Treatment (Regorafenib)
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: The 95% CIs will be calculated using the Wilson method. Will be analyzed using KM curves.
Time Frame: From start of treatment until death due to any cause, assessed up to 4 years
Population: Due to insufficient accrual (only 3 accrued), no analysis was performed.
Arm/Group | Treatment (Regorafenib)
Number analyzed (Participants) | 0

4. Secondary Outcome: Incidence of Adverse Events, Assessed According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Description: Toxicity profile will be summarized by attribution: regorafenib-related and all reported, course: course 1 and all courses, type, and grade: grade 1-2, 3-4, and 5.
Time Frame: Up to 4 years
Population: Data not collected
Arm/Group | Treatment (Regorafenib)
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Biomarkers Such as Messenger Ribonucleic Acid (mRNA) Levels or Germline Variations of Genes Related to Angiogenesis
Description: The associations between biomarkers and clinical outcomes (6-month PFS, response, PFS, and overall survival) will be analyzed in univariate analysis first using appropriate methods. Multivariable analyses will be conducted to evaluate the independent effect of a marker on clinical outcome. All tests will be two-sided at a significance level of 0.05. P values will be adjusted for multiple comparisons.
Time Frame: Up to 4 years
Population: Analysis not done. Only 3 subjects were enrolled out of the accrual goal of subjects.
Arm/Group | Treatment (Regorafenib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject received the initial study drug administration and continued throughout the study until 30 days after the last dose or until resolution of adverse event if beyond 30 days after last dose.
Description: Adverse events are assessed during regularly scheduled follow up.
Arm/Group | Treatment (Regorafenib)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Regorafenib) (N=3)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Regorafenib) (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (3)
Paronychia (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3)
Dysgeusia (Nervous system disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Hoarseness (Reproductive system and breast disorders) | 2 (2)
Voice alteration (Reproductive system and breast disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT02259725/Prot_SAP_000.pdf